CLINICAL TRIAL: NCT01712295
Title: New Formulation of Salicylate to Improve Treatment of Common Skin Warts
Brief Title: 17% Salicylate Versus 17% Salicylate-Ethyl Pyruvate for Plantar Foot Warts
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Grossman, Michael, D.P.M. (Individual)
Collaborators: Main Line Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R12-3128
Record Dates: First submitted 2012-10-19; First posted 2012-10-23 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-10

CONDITIONS: Warts
Keywords: Warts; salicylic acid; ethyl pyruvate
MeSH Terms: conditions — Warts | interventions — Salicylates; ethyl pyruvate; compound W

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 17% Salicylate with Ethyl Pyruvate (Experimental): Subjects with plantar wart(s) will apply the product to warts twice a day for up to 16 weeks.
  Interventions: Drug: 17% Salicylate with ethyl pyruvate
- 17% salicylate (Active Comparator): subjects will apply 17% salicylate (standard of care treatment) to plantar skin wart(s) twice a day for up to 16 weeks
  Interventions: Drug: Salicylates

INTERVENTIONS:
Drug: 17% Salicylate with ethyl pyruvate
  Other Names: Compound W
  Arms: 17% Salicylate with Ethyl Pyruvate
Drug: Salicylates
  Arms: 17% salicylate

SUMMARY:
Plantar warts on the sole of the foot are among the most common warts seen in podiatry clinics. Some patients are readily cured by simple standard of care treatments that include wart debridement (trimming or excision) and application of 17% salicylate (commercially known as Compound W)or by other treatments that may be painful and affect mobility. No treatment is consistently effective and most patients fail treatment multiple times.

Ethyl pyruvate (EP)is a common food additive noted to be 'generally regarded as safe' that may improve the activity of salicylate in wart treatment by improving the ability to penetrate and/or persist in the skin. The use of 17% salicylate with the addition of EP may improve cures of common foot plantar warts in subjects who also be receiving other standard-of-care treatment.

ELIGIBILITY:
Inclusion Criteria:

* evidence of skin plantar wart(s)

Exclusion Criteria:

* iodine allergy

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-12 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
To determine if salicylate with ethyl pyruvate (SA-EP) eliminates plantar warts more quickly than salicylate (SA) alone. | 16 weeks
  Subjects' wart(s) are treated with SA or SA-EP every two weeks for up to 16 weeks.

SECONDARY OUTCOMES:
To determine if salicylate with ethyl pyruvate (SA-EP) in treatment of plantar warts causes adverse events other than those known to occur with SA (salicylate)alone. | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Grossman, DPM, Principal Investigator
Locations (1):
- Main Line Foot and Ankle Center, Ardmore, Pennsylvania, United States